CLINICAL TRIAL: NCT04544384
Title: Acute Myocardial Infarction in Iceland, is There a Gender Difference in Treatment and Survival?
Status: Completed | Type: Observational
Sponsor: Landspitali University Hospital (Other)
Collaborators: Statistics Iceland (Unknown)
Responsible Party: Sponsor
Other Study IDs: LSH-19-003
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Acute Myocardial Infarction; Coronary Angiography
Keywords: Acute myocardial infarction; Gender difference; Long-term survival; Excess mortality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All patients in Iceland with STEMI (2008-2018) and NSTEMI (2013-2018) that underwent coronary angiography and had obstructive coronary artery disease were included. Information about patients and angiography results and treatment were obtained from the Swedish Coronary Angiography and Angioplasty Registry (SCAAR). Survival was estimated with Kaplan-Meier method. Cox regression analysis were used to identify significant risk factors for long-term mortality. Relative survival was defined as observed survival divided by expected survival of the population of Iceland

DETAILED DESCRIPTION:
Methods This is a retrospective observational nationwide study of all patients, aged 18 years and older, who underwent coronary angiography for acute myocardial infarction (AMI) during the study period. All procedures were performed at Landspitali University Hospital, which is a tertiary referral center and the only institution performing coronary angiographies in Iceland. The study period was from January 1, 2008 to December 31, 2018 for ST elevation myocardial infarction (STEMI and from January 1, 2013 to December 31, 2018 for non-ST elevation myocardial infarction (NSTEMI). For multiple admissions, the first was retained.

Information about patient demographics, cardiovascular risk factors, comorbidities, angiography results and treatment were obtained from the Swedish Coronary Angiography and Angioplasty Registry (SCAAR), a Swedish Web-based database also used in Iceland that prospectively record both patient- and procedure-related factors. All data are registered by the treating physician and nurses at the time of the procedure.

Clinical definitions Cases of acute myocardial were defined as STEMI and NSTEMI, according to the current European Society of Cardiology guidelines, and determined by the attending cardiologist [18]. The NSTEMI diagnosis was introduced into the database 2013 and there was also a change in the Troponin analysis used at that time. This is the reason why we chose to have a shorter study period for the NSTEMI patients. We excluded patients that had not significant coronary artery stenoses. Cardiovascular risk factors, including hypertension, diabetes mellitus, smoking status, statin use, body mass index (BMI) and renal function were recorded. Chronic kidney disease (CKD) was staged according to the Kidney Disease Outcome Quality Initiative (KDOQI) classification. Estimated glomerular filtration rate (eGFR) was calculated from serum creatinine measurements using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation, and CKD was defined as eGFR < 60 mL/min/1.73 m2 (stage 3-5).

Prior MI, percutaneous coronary intervention (PCI) and coronary artery bypass grafting (CABG) were recorded as defined in the database. Since these were AMI patients, they were all done urgently but it was also recorded whether they were done acutely as primary PCIs. The results of the coronary angiography were expressed as the number of vessels involved with significant stenoses or left main stem disease based on angiographic results. If PCI was performed, it was recorded whether patients received aspirin (acetylsalicylic acid) or adenosine diphosphate receptor (ADP) inhibitor before or during the procedure. The choice of treatment, medical therapy alone, PCI or CABG, was at the discretion of the attending interventional cardiologist and/or the heart team.

Observed and Expected Survival Data for all-cause mortality were extracted through linkage with Statistics Iceland. Patients were followed up for their vital status after hospitalization, with censoring at the end of follow-up on October 23, 2019. Expected survival was derived from the general population of Iceland matched to observed survival for the study population by sex, age and year of hospitalization.

Statistical analysis All calculations were performed using R software version 3.3.3 (R Foundation for Statistical Computing, Vienna, Austria). All continuous variables were normally distributed and were compared with Student´s t-test and presented as mean ± standard deviation (SD). Categorical variables were compared using Chi-square test if the observed data was over five, otherwise Fisher´s Exact test was performed. Statistical significance was prespecified at 5% (P < 0.05) Kaplan-Meier curve was plotted to assess the estimated long-term survival and the two groups were compared using a log-rank test. To identify independent prognostic factors for survival, a Cox multivariate analysis was used, represented as hazard ratios with 95% confidence intervals.

Relative survival was defined as the observed survival among patients with AMI divided by expected survival in populace of Iceland matched by sex, age and year.

As individual patients were not identified, obtaining individual consent for the study was not obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSTEMI during 2013-2018 that underwent coronary angiography
* Patients with STEMI during 2008-2018 that underwent coronary angiography

Exclusion Criteria:

* Normal coronary arteries on coronary angiography
* Not first presentation of NSTEMI or STEMI during the study period
* Lost survival data

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients, aged 18 years and older, who underwent coronary angiography for acute myocardial infarction (AMI) during the study period. All procedures were performed at Landspitali University Hospital, which is a tertiary referral center and the only institution performing coronary angiographies in Iceland. The study period was from January 1, 2008 to December 31, 2018 for ST elevation myocardial infarction (STEMI and from January 1, 2013 to December 31, 2018 for non-ST elevation myocardial infarction (NSTEMI).
Sampling Method: Non-Probability Sample
Enrollment: 3257 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Long-term Survival | From time of NSTEMI/STEMI to mortality or October 23, 2019
  Compare treatment and survival of men and women with NSTEMI or STEMI and obstructive coronary artery disease.

SECONDARY OUTCOMES:
Independent risk factors for mortality | For NSTEMI (2013-2018) and For STEMI (2008-2018)
  Independent risk factors for mortality are found by Cox regression analysis
Relative survival | For NSTEMI (2013-2018) and For STEMI (2008-2018)
  Defined as observed survival, among patients with STEMI and NSTEMI, divided by expected survival in the matched populace of Iceland.

CONTACTS AND LOCATIONS:
Overall Officials: Ingibjorg Gudmundsdottir, Phd, MD, Study Director — Landspitali